CLINICAL TRIAL: NCT01994408
Title: Automatic Medication Increase Protocol in the Treatment of Elevated Blood Pressure
Brief Title: Default BP Medication Intensification
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Florian Rader, MD, MSc, Assistant Professor, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00030558
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension
Keywords: physician inertia; hypertension; telemedicine; mobile technology
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: default drug escalation
Oversight: Data Monitoring Committee: No

ARMS (1):
- default intensification arm (all) (Experimental): all subjects will receive blister packs with weekly increasing blood pressure medications. There is no control arm for this study
  Interventions: Other: default intensification

INTERVENTIONS:
Other: default intensification — The investigators will determine which blood pressure medications to use. No specific drug will be tested but rather the automatic intensification of medications is the intervention. Examples of drugs used in this study are calcium channel blockers (e.g., amlodipine 2.5 mg to 10 mg) or ACE-inhibitors (e.g., lisinopril 5 mg to 40 mg) or diuretics (HCTZ 25 mg).
  Other Names: weekly increasing blood pressure medications.

SUMMARY:
High blood pressure leads to heart attacks and strokes which can be prevented by blood pressure-lowering medication. However, the current office-based prescription of one pill and one dose at a time is ineffective. the investigators want to pilot-test a more effective patient-centered treatment approach, where patients will receive a prescription with gradual but automatic weekly increases of dose and number of pills. Patients will measure their blood pressure with an iPhone compatible cuff, which transmits readings to the doctor or pharmacist, who will stop escalation when the desired blood pressure level is reached. The investigators hypothesize that the intervention will decrease the time to control blood pressure and increase the overall rate of blood pressure control. Therefore, this new treatment model could prevent heart attacks and strokes, and reduce healthcare costs.

DETAILED DESCRIPTION:
This is a pilot 2A trial of an innovative behavioral economics theory-based antidote for physician inertia in the medical treatment of hypertension (HTN). In the current reactive physician-centered model, blood pressure (BP) is measured and medical decisions are made in the physician office; when deciding whether or not to prescribe new medication for a high office BP reading, the physician's default behavior is inaction. The investigators propose default medication intensification as a new patient-centered/pharmacist-assisted proactive treatment model to eliminate physician inertia. For enrolled patients with office BP>155/95, the physician will prescribe a one-month protocol that automatically escalates drug dose and drug number each week. The pharmacist will fill the prescription in a blister pack to simplify adherence. The patient will measure daily home BP with an iPhone cuff that transmits the data electronically to the pharmacist, who will halt the protocol if goal home BP<135/85 is achieved ahead of schedule. the investigators will pilot test the feasibility and safety of self-monitoring plus the new automatic intensification protocol packaged in blisters. Default medication intensification could revolutionize HTN treatment and reduce healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years old
* office BP of ≥160 mmHg systolic and ≥100 mmHg diastolic (treated or untreated) AND <180 mmHg systolic.

Exclusion Criteria:

* chronic kidney disease
* symptomatic coronary artery disease
* congestive heart failure
* more than mild valvular heart disease
* Diabetes mellitus
* obstructive left ventricular hypertrophy
* severe electrolyte abnormalities
* multiple medication intolerances
* orthostatic hypotension
* cognitive impairment and mental disorders affecting ability to self-monitor BP
* patients who are unwilling to measure and transmit BP readings throughout the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Symptomatic hypotension | from enrollment to 12 weeks
  Primary safety outcome is symptomatic hypotension during study participation (12 weeks). Safety monitoring will be achieved with patient-directed iPhone-based BP measuring and transmitting to study staff.

SECONDARY OUTCOMES:
hypertension control rate | at 12 weeks
  The investigators will assess blood pressure throughout the study period (12 weeks) with iPhone based technology. Hypertension control is defined as home blood pressure <135/85 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Florian Rader, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Phillips LS, Branch WT, Cook CB, Doyle JP, El-Kebbi IM, Gallina DL, Miller CD, Ziemer DC, Barnes CS. Clinical inertia. Ann Intern Med. 2001 Nov 6;135(9):825-34. doi: 10.7326/0003-4819-135-9-200111060-00012. PMID 11694107
- [Background] O'Connor PJ. Overcome clinical inertia to control systolic blood pressure. Arch Intern Med. 2003 Dec 8-22;163(22):2677-8. doi: 10.1001/archinte.163.22.2677. No abstract available. PMID 14662620
- [Background] Green BB, Cook AJ, Ralston JD, Fishman PA, Catz SL, Carlson J, Carrell D, Tyll L, Larson EB, Thompson RS. Effectiveness of home blood pressure monitoring, Web communication, and pharmacist care on hypertension control: a randomized controlled trial. JAMA. 2008 Jun 25;299(24):2857-67. doi: 10.1001/jama.299.24.2857. PMID 18577730
- [Background] Bray EP, Holder R, Mant J, McManus RJ. Does self-monitoring reduce blood pressure? Meta-analysis with meta-regression of randomized controlled trials. Ann Med. 2010 Jul;42(5):371-86. doi: 10.3109/07853890.2010.489567. PMID 20504241